CLINICAL TRIAL: NCT02214563
Title: Cholecalciferol Supplementation for Anemia and Mineral and Bone Disorder in Hemodialysis Patients (CHAMBER): A Multicenter, Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Cholecalciferol Supplementation for Anemia and Mineral and Bone Disorder in Hemodialysis Patients
Acronym: CHAMBER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takayuki Hamano (Other)
Collaborators: The Japan Kidney Foundation (Other); Molecular Physiological Chemistry Laboratory, Inc. (Other); Obi clinic (Unknown); Higashikouri Hospital (Unknown); Nishi clinic (Unknown); Futaba clinic (Unknown); Akebono clinic (Unknown)
Responsible Party: Sponsor-Investigator, Takayuki Hamano, Associate Professor, Osaka University
Organization: Osaka University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CKDR-003
Record Dates: First submitted 2014-08-10; First posted 2014-08-12 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Kidney Failure, Chronic; Anemia; Vitamin D Deficiency; Bone Diseases, Metabolic
Keywords: Vitamin D; Cholecalciferol; Hepcidins; Renal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia; Vitamin D Deficiency; Bone Diseases, Metabolic | interventions — Cholecalciferol; Vitamin D; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Thrice-weekly cholecalciferol (Active Comparator): Capsule containing 3,000 IU of cholecalciferol will be given at the end of each hemodialysis session. Dissolved with olive oil and coated by soft capsule made of gelatin and glycerin.
  Interventions: Dietary Supplement: Cholecalciferol
- Monthly cholecalciferol (Active Comparator): Capsules containing a dose equivalent to 9,000 IU/week will be given at the end of the first hemodialysis session in the 3rd week of each month. Dissolved with olive oil and coated by soft capsule made of gelatin and glycerin.
  Interventions: Dietary Supplement: Cholecalciferol
- Thrice-weekly placebo (Placebo Comparator): Olive oil coated by soft capsule made of gelatin and glycerin.
  Interventions: Dietary Supplement: Olive oil
- Monthly placebo (Placebo Comparator): Olive oil coated by soft capsule made of gelatin and glycerin.
  Interventions: Dietary Supplement: Olive oil

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Made for this trial by Molecular Physiological Chemistry Laboratory, Inc.
  Other Names: vitamin D; vitamin D3
  Arms: Monthly cholecalciferol; Thrice-weekly cholecalciferol
Dietary Supplement: Olive oil
  Arms: Monthly placebo; Thrice-weekly placebo

SUMMARY:
The purpose of this study is to determine whether cholecalciferol supplementation decrease the blood concentrations of hepcidin-25 in hemodialysis patients.

DETAILED DESCRIPTION:
There are 4 arms in this study: (1) Thrice-weekly cholecalciferol supplementation (3,000 IU), (2) Monthly cholecalciferol supplementation (equivalent to 9,000/week), (3) Thrice-weekly placebo, and (4) Monthly placebo. The primary analyses will be done regarding 2 cholecalciferol groups and 2 placebo groups as one group each, and we will evaluate the effect of cholecalciferol regardless of the supplementation regimen. As the secondary analyses, we will examine if there is any difference between thrice-weekly and once-monthly supplementation regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage renal disease receiving thrice-weekly maintenance hemodialysis
* On treatment with erythropoietin stimulating agent
* With written informed consent

Exclusion Criteria:

* On treatment with epoetin beta pegol as ESA
* On supplementation with native vitamin D
* Hypercalcemia (>=10.5 mg/dL of corrected serum calcium)
* On treatment with intravenous iron agents
* Judged as ineligible to the randomized study by the investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of hepcidin-25 | The 3rd month
Serum concentrations of hepcidin-25 | The 3rd day

SECONDARY OUTCOMES:
Serum concentrations of hepcidin-25 | The 6th month
Percent change of erythropoietin resistance index (ERI) overtime | Up to the 6th month
  ERI = Average weekly dose of erythropoiesis-stimulating agents (ESA) over prior 4 weeks / post-dialysis body weight (kg) / Hb (g/dL)
Blood concentrations of 1,25-dihydroxyvitamin D, bone specific alkaline phosphatase (BAP), and tartrate-resistant acid phosphatase (TRAcP) 5b | The 3rd month
  In the secondary analysis, we will adjust baseline concentrations when comparing the groups.
Blood concentrations of 1,25-dihydroxyvitamin D, bone specific alkaline phosphatase (BAP), and tartrate-resistant acid phosphatase (TRAcP) 5b | The 6th month
  In the secondary analysis, we will adjust baseline concentrations when comparing the groups.
Blood concentrations of high-sensitive C reactive protein (CRP), interleukin (IL)-6, and tumor necrosis factor (TNF)-alpha | The 3rd day
  In the secondary analysis, we will adjust baseline concentrations when comparing the groups.
Blood concentrations of high-sensitive C reactive protein (CRP), interleukin (IL)-6, and tumor necrosis factor (TNF)-alpha | The 3rd month
  In the secondary analysis, we will adjust baseline concentrations when comparing the groups.
Blood concentrations of high-sensitive C reactive protein (CRP), interleukin (IL)-6, and tumor necrosis factor (TNF)-alpha | The 6th month
  In the secondary analysis, we will adjust baseline concentrations when comparing the groups.
Blood concentrations of calcium, phosphate, and intact parathyroid hormone overtime | Up to the 6th month
  In the secondary analysis, we will adjust baseline concentrations when comparing the groups.

OTHER OUTCOMES:
Hypercalcemia | Up to the 6th month
  >=10.5 mg/dL of albumin corrected calcium

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiharu Tsubakihara, MD, PhD, Study Chair — Department of Comprehensive Kidney Disease Research, Osaka University Graduate School of Medicine
Locations (7):
- Japan (7):
  - Hyogo Prefectural Nishinomiya Hospital, Nishinomiya, Hyōgo
  - Higashikouri hospital, Hirakata, Osaka
  - Department of Comprehensive Kidney Disease Research, Osaka University Graduate School of Medicine, Suita, Osaka
  - Akebono clinic, Kumamoto
  - Obi clinic, Osaka
  - Nishi clinic, Osaka
  - Futaba clinic, Osaka

REFERENCES:
- [Derived] Obi Y, Yamaguchi S, Hamano T, Sakaguchi Y, Shimomura A, Namba-Hamano T, Mikami S, Nishi O, Tanaka M, Kamoto A, Obi Y, Tomosugi N, Tsubakihara Y, Isaka Y. Effect of cholecalciferol on serum hepcidin and parameters of anaemia and CKD-MBD among haemodialysis patients: a randomized clinical trial. Sci Rep. 2020 Sep 23;10(1):15500. doi: 10.1038/s41598-020-72385-w. PMID 32968158
- See also: Link to the report which showed the negative effect of vitamin D on blood hepcidin-25 concentration in human subjects — http://www.ncbi.nlm.nih.gov/pubmed/24204002